CLINICAL TRIAL: NCT05038956
Title: Serum Bupivacaine Concentration Levels After Intermittent Bolus Injections Through Erector Spinae Plane Peripheral Catheter
Brief Title: Serum Bupivacaine Concentration Levels After Intermittent Bolus Injections Via Erector Spinae Plane Peripheral Catheter
Status: Withdrawn | Type: Observational
Why Stopped: No immediate plans to start the study. Issues with testing materials.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kasinda Goodwin, Assistant Professor (Clinical), University of Utah
Other Study IDs: IRB 00142099
Record Dates: First submitted 2021-08-03; First posted 2021-09-09 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-07

CONDITIONS: Video-assisted Thoracic Surgery (VATS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Each participant will have 5 mL of venous blood drawn to assess serum bupivacaine levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate the serum bupivacaine concentrations over time after 0.125% bupivacaine is deposited every 6 hours in the erector spinae plane in patients who undergo unilateral VATS.

DETAILED DESCRIPTION:
Pain control is an important aspect of recovery for patients who undergo thoracic surgery. Over the past several decades, thoracic surgery has shifted from open thoracotomies to video-assisted thoracic surgery (VATS) with the result of less morbidity, fewer postoperative complications and less postoperative pain compared to open thoracic procedures. However, postoperative acute and chronic thoracic pain remain a main clinical issue with VATS and contributes to patient suffering as well as the ability to meet early rehabilitation goals. Chest wall pain has traditionally been managed with epidural analgesia and/or by narcotic medication administration (such as morphine, hydromorphone and oxycodone). These modalities, however, carry a high risk of serious effects such as epidural hematomas, dural puncture, pneumothorax, hypotension, infection as well as cough suppression, constipation, drowsiness and mental status changes. Additionally, patients who are on anticoagulants or antiplatelet therapy may not be eligible for epidural analgesia. Furthermore, the short- and long-term analgesic benefits of epidural analgesia has been shown to be inconsistent in the setting of VATS.

A relatively new technique used for post-operative pain control in thoracic surgery is the use of fascial plane blocks, specifically the erector spinae plane block (ESPB). The ESPB was first described in 2016 by Forero et al. in 4 case reports: 2 patients with chronic thoracic neuropathic pain and 2 patients with acute postoperative chest wall pain 8. Since that time the ESPB has been widely adopted as a regional technique used in thoracic, breast, abdominal and lumbar surgery. This block is achieved by depositing long-acting local anesthetic medication in the fascial plane deep to the erector spinae muscles and superficial to the transverse process, to achieve a distribution along several vertebral rami of the spinal nerves and intercostal spaces. Radiographic evidence suggests that local anesthetic injected at the ESP spreads both cranially and caudally as the plane is continuous along the vertebral column. These rami carry visceral motor, somatic motor and sensory information to and from the skin and deep muscles of the back.

In thoracic surgery, the ESPB has shown to decrease opioid consumption and pain scores in patients who undergo VATS within the first 24 hours when compared to no block and also when compared to other fascial plane blocks such as the serratus plane block. In the literature thus far, complications are rare.

Although the literature has quickly grown regarding erector spinae blocks over the last four years, specific information regarding dosing regimens for both single injection and intermittent bolus dosing through an erector spinae catheter remains limited. Most of the current information from the erector spinae block lies in case reports. In reviews of the current practices, it appears that ropivacaine and bupivacaine are the most commonly used local anesthetics with injection volumes ranging from 20 mL to 40 mL and concentrations ranging from 0.25%-0.5%. Most case reports describe single injection, while approximately 20% describe dosing either intermittently or continuously through a catheter. It is thought that because this block is a fascial plane block its' success depends, in part, on the volume and concentration of local anesthetic injected in the erector spinae plane to achieve maximal craniocaudal dermatomal distribution. It is in these scenarios that clinicians must balance achieving maximal analgesic benefit from this block with safety concerns for local anesthetic systemic toxicity (LAST).

There are no documented cases described of a patient experiencing LAST from an erector spinae block or erector spinae nerve catheter, however there is some information regarding the safety of similar fascial plane blocks. Convulsions following bilateral ultrasound guided transversus abdominis plane blocks following cesarean analgesia have been described. Trabelsi et al. describe the pharmacokinetics of bupivacaine after bilateral transversus abdominis plane blocks and found that mean peak serum bupivacaine concentrations was 30 minutes from the time of injection. However, during this study, three subjects had serum bupivacaine concentrations above the quoted toxic threshold. Furthermore, data analyzing serum concentration of local anesthetic overtime through the use of catheters is also lacking. In a study of pediatric patients with continuous paravertebral infusions it was found that serum concentration of bupivacaine was >3 mcg/mL in several infants at 30-48 hours. These studies emphasize the need for better understanding local anesthetic uptake from fascial planes blocks.

In prior studies that have attempted to illustrate the pharmacokinetics of local anesthetic uptake to serum concentrations, data has been scattered to such a degree that the investigators cannot accurately extrapolate trends. A previous study at our institution measured serum ropivacaine levels following local infiltration in the knee joint and found max serum concentrations ranging from 4 to 24 hours. In an observational study examining the pharmacokinetics of liposomal bupivacaine placed in the intercostal space, maximal serum levels ranged from 15 minutes to 48 hours. In a study analyzing the pharmacokinetics of bupivacaine following bilateral transversus abdominis plane blocks, all individual peak plasma levels were recorded between 10 and 90 minutes. With this proposed observational study, the investigators expect to see scattered data which is why the need for such tight time intervals of measurements and the amount of measurements. Besides looking at the maximum serum concentration of bupivacaine following the boluses, an additional important aspect of this observational study is to see if there is a stacking effect of plasma bupivacaine levels following repeated dosing through the catheter. Taketa et al, examined serum levels following continuous infusions of local anesthetic in the paravertebral and erector spinae planes and found building serum levels with the continuous infusion. There have been no studies to analyze if there is a stacking effect of local anesthetic in serum levels following multiple intermittent bolus doses.

Currently, no publication exists that report serum bupivacaine concentration over time following initial bolus in the erector spinae plane or following intermittent boluses of erector spinae plane catheters. This information is important to ensure that safe serum bupivacaine concentrations are maintained when considering optimal bolus dosing and intervals for erector spinae plane catheters. The current practice at the University of Utah is to bolus 25 mg of bupivacaine hydrochloride (HCL) (20 mL of 0.125% bupivacaine) through erector spinae catheters every six hours. Occasionally this regimen is ineffective and the investigators consider increasing the concentration, volume or decreasing the interval of bupivacaine administration in order to obtain better postoperative analgesia. However, increasing bupivacaine dosing also increases the risk of local anesthetic toxicity. Striking the appropriate balance between safety and maximally effective postoperative analgesia has been clinically challenging for our regional anesthesiologists and for subject experts across the world. There are no consensus data on the effective-safe dosing of these catheters. Having this knowledge will help ensure a safe practice of local anesthetic usage for unilateral thoracic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* having a unilateral video assisted thorascopic surgery who have preoperative placement of an erector spinae plane catheter.

Exclusion Criteria:

* Known hepatic dysfunction or renal insufficiency (creatinine >1.5 mg/dL)
* allergy to the study medication
* pregnancy
* incarceration
* inability to communicate with the investigators
* morbid obesity (body mass index >40 mg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are having unilateral video assisted thorascopic surgery at the University of Utah or Huntsman Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in pharmacokinetics of bupivacaine placed in the erector spinae plane between 6 time points | 30, 60, 90, 120, 240 and 360 minutes following the initial, 2nd and 5th boluses.
  Each participant will have 5 mL of venous blood drawn to assess serum bupivacaine levels

SECONDARY OUTCOMES:
Change in stacking effect of plasma bupivacaine levels between 6 time points | 30, 60, 90, 120, 240 and 360 minutes following the initial, 2nd and 5th boluses.
  Each participant will have 5 mL of venous blood drawn

CONTACTS AND LOCATIONS:
Overall Officials: Kasinda Goodwin, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States